



## PARTICIPANT CONSENT FORM (MAIN STUDY)

Title of Project: Digital Assessment of Wellbeing in New Parents (DAWN-P) app use phase

| | Activities | Initials |
|---|---|---|
| 1 | I confirm that I have read the attached information sheet (Version X, date XX/XX/XXXX) for the above study and have had the opportunity to consider the information and ask questions and had these answered satisfactorily. | |
| 2 | I understand that my participation in the study is voluntary and that I am free to withdraw at any time without giving a reason and without detriment to myself. I understand that it will not be possible to remove my data from the project once it has been anonymised and forms part of the data set. I agree to take part on this basis. | |
| 3 | I agree to my GP being informed of my participation in the study | |
| 4 | I agree that any data collected may be published in anonymous form in academic books, reports or journals. | |
| 5 | I understand that there may be instances where, during the course of the study, information is revealed which means that the researchers will be obliged to break confidentiality and this has been explained in more detail in the information sheet. | |
| 6 | Participating perinatal women: I understand that relevant sections of my medical notes may be looked at by the researchers. I give permission for these individuals to have access to my records. | |
| | I understand that data collected during the study and sections of my medical notes may be looked at by individuals from The University of Manchester, Manchester University Foundation NHS Trust or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to this information. | |
| | Participating partners: I understand that data collected during the study may be looked at by individuals from The University of Manchester, Manchester University Foundation NHS Trust or regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to this information. | |
| 7 | I agree to take part in this study. | |

Data Protection: The personal information we collect and use to conduct this research will be processed in accordance with data protection law as explained in the Participant Information Sheet and the Privacy Notice for Research Participants (http://documents.manchester.ac.uk/display.aspx?DocID=37095).

| Name of participant | <br>Date | Signature |
|-------------------------------|----------|-----------|
| Name of person taking consent | Date | Signature |

## **Optional additional consent:**

| 8 | I agree that the researchers may contact me in future about other research projects. |
|---|---|
| 9 | I agree that the researchers may retain my contact details in order to provide me with a summary of the findings for this study. |

Data Protection: The personal information we collect and use to conduct this research will be processed in accordance with data protection law as explained in the Participant Information Sheet and the Privacy Notice for Research Participants (http://documents.manchester.ac.uk/display.aspx?DocID=37095).

| Name of participant | Date | Signature |
|-------------------------------|----------|-----------|
| Name of person taking consent | <br>Date | Signature |